CLINICAL TRIAL: NCT04486872
Title: A Single-arm, Open-label, Dose Escalation Study to Explore Safety, Efficacy and Pharmacokinetics of Autologous Humanized Anti-CD19 and Anti-CD20 Dual Specific CAR-T Cells in Adult Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma
Brief Title: An Exploratory Clinical Trial of Autologous Humanized Anti-cluster of Differentiation Antigen 19/20(CD19/CD20) Dual Specific CAR-T Cells Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, shentu jianzhong, Prof, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-02 POC-01
Record Dates: First submitted 2020-07-17; First posted 2020-07-27 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 and anti-CD20 dual specific CAR-T Cells (Experimental)
  Interventions: Biological: Autologous humanized anti-CD19 and anti-CD20 dual specific CAR-T Cells

INTERVENTIONS:
Biological: Autologous humanized anti-CD19 and anti-CD20 dual specific CAR-T Cells — Autologous Humanized Anti-CD19 and Anti-CD20 Dual Specific CAR-T Cells injection. Within 3 to 5 days after the pretreatment, the subjects received a single A-02 reinfusion, the infusion dose of each group of subjects 1.00 × 10^6/kg, 3.00 × 10^6/kg or 5.00 × 10^6/kg (if applicable), it is recommended to complete the infusion within 30 min after cell recovery.

SUMMARY:
This is a single-arm, open-label, dose escalation, phase I study, aiming to evaluate the safety and efficacy of Autologous Humanized Anti-CD19 and Anti-CD20 Dual Specific Chimeric Antigen Receptor (CAR) T-cells in patient with relapsed or refractory diffuse B cell lymphoma.

DETAILED DESCRIPTION:
CD19 CAR-T cell therapy has made breakthroughs in the treatment of B cell lymphoma and leukemia, but 30% of patients still have antigen escape, which may be related to variants in tumor cells and the expansion of CD19-negative tumor cells after treatment with CD19 CAR-T cells. CD19/CD20 bispecific CAR-T cell targeting multiple antigens can attack tumor cells while overcoming tumor antigen escape caused by a single target, maximizing efficacy and duration of treatment, and can also solve the problem of uneven distribution or low expression of single target on the tumor surface.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or her/his legally guardian(s) must sign the informed consent form approved by the Institutional Ethics Committee (IEC) prior to any screening procedures;
2. Subjects aged 18 years or older with relapsed or refractory DLBCL (including primary mediastinal large B-cell lymphoma and transformed follicular lymphoma), of which refractory is defined as:

   * Have no response to the recent treatment including:

     * The best response to the treatment regimen is progressive disease (PD) ,or;
     * stable disease(SD) which maintained less than 6 months after the last treatment, or;
   * not suitable for autologous hematopoietic stem cell transplantation (ASCT), or ASCT refractory, including:

     * progressive disease after ASCT or relapse within 12 months (relapse must be confirmed by biopsy), or;
     * If remedial treatment is given after ASCT, the subject must have no response or relapse after the last treatment.
3. Subjects who have previously received ≥2 lines treatment, and at least including:

   * Anti-CD20 monoclonal antibody(rituximab), unless the CD20 negative;
   * A chemotherapy regimen containing anthracyclines;
   * The DLBCL patients who transformed from follicular lymphoma must have previously received chemotherapy for follicular lymphoma and have developed chemotherapy-refractory diseases after transform to DLBCL.
4. Confirmation for either CD19 or CD20 positivity using immunohistochemistry or flow cytometry(accepting the previous results from the a third-level grade A hospitals before the collection of peripheral blood mononuclear cells or peripheral blood. For CD20 positive only, the investigator needs to determine whether the treatment benefit);
5. According to the preliminary assessment of Hodgkin's lymphoma and non-Hodgkin's lymphoma, staging and response assessment recommendations (2014 version), there is at least one measurable lesion at baseline;
6. If the subject has received a single target in the past, such as CD19-CAR cell therapy, it must be confirmed that the disease has progressed or relapsed after treatment and is at least 1 month from the planned single collection period
7. Life expectancy ≥12 weeks;
8. Eastern Cooperative Oncology Group (ECOG) performance status that is either 0 or 1 at screening;
9. Adequate organ function:

   * Renal function defined as:

     * A serum creatinine of ≤1.5 × Upper Limit of Normal(ULN), or;
     * Estimated Glomerular Filtration Rate (eGFR) ≥60 ml/min/1.73m2；[eGFR=186×（age）-0.203×SCr-1.154（mg/dl）， female ×0.742 on the basis of the calculation results]；
   * Liver function defined as:

     * Alanine aminotransferase (ALT)≤ 5 × Upper Limit of Normal(ULN) for age, and;
     * Total bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert-Meulengracht syndrome; patients with Gilbert-Meulengracht syndrome may be included if their total bilirubin is ≤ 3.0 × ULN and direct bilirubin ≤ 1.5 × ULN.
   * Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and blood oxygen saturation > 91% on room air;
10. Hemodynamically stable and Left Ventricle Ejection Fraction (LVEF) ≥ 45% confirmed by echocardiogram or Multigated Radionuclide Angiography (MUGA);
11. Adequate bone marrow reserve without transfusions defined as:

    * Absolute neutrophil count (ANC) >1×10^9 /L；
    * Absolute lymphocyte count (ALC) ≥0.3×10^9 /L；
    * Platelets ≥50×10^9 /L;
    * Hemoglobin > 8.0 g/dl;
12. Subjects who use the following drugs should meet the following criteria:

    * Steroids: Therapeutic doses of steroids must be stopped 2 weeks prior to A-02 infusion. However, the following physiological replacement doses of steroids are allowed: < 6 - 12 mg/m2/day hydrocortisone or equivalent;
    * Immunosuppression: Any immunosuppressive medication must be stopped ≥ 4 weeks prior to sign the informed consent form;
    * Anti-proliferative therapy other than pretreatment chemotherapy within 2 weeks of A-02 infusion;
    * CD20 antibody-related treatment must be discontinued within 4 weeks of A-02 infusion or 5 half-lives (whichever is longer);
    * CNS disease prophylaxis must be stopped > 1 week prior to A-02 infusion (e.g. intrathecal methotrexate);
13. The investigator judged that the subject recovered from the toxicity of the previous anti-tumor treatment to grade 1 or below (except for special grade 2 or below toxicity that cannot be recovered in a short period of time, such as hair loss), suitable for pretreatment. Chemotherapy and treatment of CAR-T cells;
14. Women of child-bearing potential and all male subjects must agree to use highly effective methods of contraception for at least 12 months following A-02 infusion and until CAR-T cells are no longer present by Polymerase chain reaction(PCR) on two consecutive tests.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be enrolled:

1. Subjects who have received any CD19/CD20 dual-target cell therapy products before signing the informed consent form;
2. Subjects with detectable cerebrospinal fluid malignant cells or brain metastases, or with a history of central nervous system (CNS) lymphoma or primary CNS lymphoma;
3. Subjects with current or previous history of central nervous system disease, such as seizures, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the central nervous system;
4. Subjects who have previously received allogeneic hematopoietic stem cell transplantation (HSCT); or suitable and consenting to Autologous hematopoietic stem cell transplantation (ASCT);
5. Chemotherapy other than lymphodepleting chemotherapy within 2 weeks of A-02 infusion;
6. Investigational medicinal product within the last 30 days prior to sign the informed consent form;
7. Subjects with active hepatitis B（defined as hepatitis B surface antigen positive, or hepatitis B core antibody positive with hepatitis B virus DNA detection value > 1000 copies/ml）or hepatitis C(HCV RNA positive);
8. Subjects positive for HIV antibody or treponema pallidum antibody;
9. Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to A-02 infusion);
10. Unstable angina and/or myocardial infarction within 6 months prior to sign the informed consent form;
11. Previous or concurrent malignancy with the following exceptions:

    * Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to sign the informed consent form);
    * In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to sign the informed consent form;
    * A primary malignancy which has been completely resected and in complete remission for ≥ 5 years;
12. Pregnant or nursing women (women of childbearing age were tested positive for pregnancy during screening period);
13. Subjects with active neurological auto immune or inflammatory disorders (e.g. Guillain Barre Syndrome, Amyotrophic Lateral Sclerosis);
14. Other conditions that the investigator thinks he/she should not be included in this clinical trial, such as poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-07-25 (Actual); Primary Completion 2022-05-11 (Estimated); Study Completion 2022-06-25 (Estimated)

PRIMARY OUTCOMES:
The types and Incidence of adverse events | Up to 12 months
  Adverse events at each visit with the NCI CTCAE v5.0 used as a guide for the grading of severity.

SECONDARY OUTCOMES:
Duration of overall response | Up to 12 months
  Time from the first occurrence of CR (complete response) or PR (partial response) to the first diagnosis of PD (progressive disease)or recurrence.
Overall survival | Up to 12 months
  Time from randomization to death due to any cause
Progression-free survival | Up to 12 months
  Time from enrollment to tumor progression or death.
Objective response rate | Up to 12 months
  The proportion of CR (complete response) and PR (partial response).
Duration of response | Up to 12 months
  Duration of response is defined as the time from the date of first occurrence of CR (complete response) or PR (partial response) to the date of the first documented PD (progressive disease) or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338